CLINICAL TRIAL: NCT01290718
Title: Study of Trastuzumab Combined With Capecitabine on HER2-positive Metastatic Breast Cancer Patients Pretreated With Trastuzumab and Taxanes or HER2- Positive Breast Cancer Patients Relapsed From (Neo)Adjuvant Therapy of Trastuzumab and Taxanes
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With Xeloda (Capecitabine) in Patients With Metastatic or Recurrent HER2-positive Breast Cancer After First-Line or (Neo)Adjuvant Therapy.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21833
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Trastuzumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 900mg/m2 bid po on days 1-14 of each 3-week cycle
Drug: trastuzumab [Herceptin] — 8mg/kg iv on day 1 of the first 3-week cycle, followed by 6mg/kg iv every 3 weeks

SUMMARY:
This single arm. open-label study will assess the efficacy and safety of Herceptin (trastuzumab) in combination with Xeloda (capecitabine) in patients with metastatic or recurrent HER2-positive breast cancer, refractory to or relapsing after chemotherapy with Herceptin and taxanes. Patients will receive Xeloda 900mg/m2 twice daily orally on days 1-14 of each 3-week cycle and Herceptin 8mg/kg intravenously (iv) on day 1 of the first cycle followed by 6mg/kg iv every 3 weeks. The anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18-65 years of age
* Histologically confirmed HER2-positive breast cancer with measurable lesions (according to RECIST criteria)
* Metastatic disease after first-line therapy or recurrent disease after (neo)adjuvant therapy with Herceptin and taxanes
* ECOG performance status 0-2

Exclusion Criteria:

* CNS metastases which are not well controlled
* Simultaneous treatment with sorivudine
* History of another malignancy within the last 5 years except for cured basal cell carcinoma of the skin and cured carcinoma in-situ of the uterine cervix
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Taiwan (3):
  - Chai Yi
  - Kaohsiung City
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine Plus (+) Trastuzumab: Participants received capecitabine 900 milligrams per square meter (mg/m^2) orally, twice daily on Days 1 to 14 followed by a 7 day rest period each 3-week cycle, along with trastuzumab 8 milligrams per kilogram (mg/kg) intravenously (iv) on Day 1 of the first 3-week cycle, followed by 6 mg/kg iv once every 3 weeks until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Capecitabine Plus (+) Trastuzumab
Started | 4
Completed | 0
Not Completed | 4
Not completed — Early termination of the study | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Capecitabine + Trastuzumab: Participants received capecitabine 900 mg/m^2 orally, twice daily on Days 1 to 14 followed by a 7 day rest period each 3-week cycle, along with trastuzumab 8 mg/kg iv on Day 1 of the first 3-week cycle, followed by 6 mg/kg iv once every 3 weeks until progressive disease or unacceptable toxicity.
Arm/Group | Capecitabine + Trastuzumab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.75 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: The tumor response was measured according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria (Version 1.1).
Time Frame: Baseline and Day 1 of Cycles 4 and 8 and every 3 weeks until unacceptable toxicity or Death
Population: Data were not analyzed due to early termination of the study.
Arm/Group | Capecitabine + Trastuzumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Disease Progression
Description: Tumor response was evaluated according to RECIST criteria (version 1.1). Progressive Disease was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Time to progression is the time from the date of first dose of drug administration to the date when first disease progression is recorded.
Time Frame: Baseline and Day 1 of Cycles 4 and 8 and every 3 weeks until unacceptable toxicity or Death
Population: Data were not analyzed due to early termination of the study.
Arm/Group | Capecitabine + Trastuzumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the time from the date of randomization to the date of death irrespective of the cause of death.
Time Frame: Baseline and Day 1 of Cycles 4 and 8 and every 3 weeks until unacceptable toxicity or Death
Population: Data were not analyzed due to early termination of the study.
Arm/Group | Capecitabine + Trastuzumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival
Description: Tumor response was evaluated according to RECIST criteria (version 1.1). Progressive Disease was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Participants without progression were censored at the date of last tumor assessment when non progression was documented.
Time Frame: Baseline and Day 1 of Cycles 4 and 8 and every 3 weeks until unacceptable toxicity or Death
Population: Data were not analyzed due to early termination of the study.
Arm/Group | Capecitabine + Trastuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) occurring up to 28 days after the last dose of study medication were to be reported.
Arm/Group | Capecitabine + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.